CLINICAL TRIAL: NCT03789812
Title: Efficacy of Different Methods of Teeth Cleaning on Oral Hygiene in Patients With Orthodontic Fixed Appliances
Brief Title: Oral Hygiene in Patients With Orthodontic Fixed Appliances
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riyadh Colleges of Dentistry and Pharmacy (Other)
Responsible Party: Principal Investigator, Omar Alkadhi, Assistant professor, Riyadh Colleges of Dentistry and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: REU/Proposal2018
Record Dates: First submitted 2018-12-27; First posted 2018-12-31 (Actual); Last update posted 2018-12-31 (Actual); Status verified 2018-12

CONDITIONS: Oral Hygiene

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Manual Toothbrush with Superfloss (Active Comparator): Patients in this group will receive Manual Toothbrush (Oral B) and Superfloss (Oral B) and will be instructed to use them three times a day.
  Interventions: Device: Manual toothbrush; Device: Superfloss
- Electric Toothbrush with Superfloss (Experimental): Patients in this group will receive Electric Toothbrush (JETPIK) and Superfloss (Oral B) and will be instructed to use them three times a day.
  Interventions: Device: Electric Toothbrush; Device: Superfloss
- Manual Toothbrush with Water Flosser (Experimental): Patient in this group will receive Manual Toothbrush and Dental Water Jet and will be instructed to use them three times a day.
  Interventions: Device: Manual toothbrush; Device: Dental Water Jet
- Electric Toothbrush with Water Flosser (Experimental): Patient in this group will receive Electric tooth brush (JETPIK) and water flosser and will be instructed to use them three times a day.
  Interventions: Device: Electric Toothbrush; Device: Dental Water Jet

INTERVENTIONS:
Device: Manual toothbrush — Soft manual toothbrush (Oral B) will be used to brush occlusal, buccal and lingual teeth surfaces.
  Arms: Manual Toothbrush with Superfloss; Manual Toothbrush with Water Flosser
Device: Electric Toothbrush — Electric toothbrush (Jetpik JP210) will be used to brush occlusal, buccal and lingual teeth surfaces.
  Arms: Electric Toothbrush with Superfloss; Electric Toothbrush with Water Flosser
Device: Superfloss — Superfloss (Oral B) will be used to clean interproximal teeth surfaces.
  Arms: Electric Toothbrush with Superfloss; Manual Toothbrush with Superfloss
Device: Dental Water Jet — Dental water jet (Jetpik JP210) will be used to clean interproximal teeth surfaces.
  Arms: Electric Toothbrush with Water Flosser; Manual Toothbrush with Water Flosser

SUMMARY:
The study aims to compare the efficacy of the use of different methods of teeth cleaning on the oral hygiene in patients with orthodontic fixed appliance

DETAILED DESCRIPTION:
Subjects were randomized into four groups, the first group will receive manual tooth brush with super floss, the second group will receive electric tooth brush with super floss, the third group will receive manual tooth brush with water dental flosser and the fourth group will receive electric tooth brush with water flosser.

ELIGIBILITY:
Inclusion Criteria:

1. participants with fixed orthodontic appliance.
2. participants age 14 years and above and didn't have mental of physical disabilities.
3. participants willing to comply with given oral hygiene instructions.

Exclusion Criteria:

1. patients with mental retardation.
2. patients with systematic diseases.

Ages: 14 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-12-03 (Actual); Primary Completion 2019-05-30 (Estimated); Study Completion 2019-07-15 (Estimated)

PRIMARY OUTCOMES:
Change in plaque index | baseline, after 4 weeks and after 8 weeks
  plaque index: 0 no plaque, 1 plaque seen only on tip of explorer or with disclosing agents, 2 plaque seen with naked eye, 3 abundance of plaque
Change in gingival index | baseline, after 4 weeks and after 8 weeks
  gingival index: 0, normal gingiva, 1 mild inflammation- slight change in color, slight edema and bleeding on probing. 2 moderate inflammation - redness, edema and bleeding on probing. 3, sever inflammation - redness, edema, and tendency to spontaneous bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- Omar AlKadhi, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No